CLINICAL TRIAL: NCT05174273
Title: Understanding the Neurocognitive Effects of Fecal Microbiota Transplantation in Major Depressive Disorder Patients With and Without Irritable Bowel Syndrome
Brief Title: Neurocognitive Effects of FMT in MDD Patients With and Without IBS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valerie Taylor (Other)
Responsible Party: Sponsor-Investigator, Valerie Taylor, Professor, Department Head, Psychiatry department, University of Calgary
Organization: University of Calgary (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IMA-FMT-MDD/IBS-2020
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder; Irritable Bowel Syndrome
Keywords: Major depression; IBS; Fecal microbiota Transplantation; Gut; Microbiome; fMRI
MeSH Terms: conditions — Depressive Disorder, Major; Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This study is a phase 2/3 open-label controlled trial (CT) in which adults with MDD with and without IBS who are being treated with an approved antidepressant medication will be assigned to additionally receive either FMT or to continue with their current treatment in a treatment as usual (TAU) arm. An IBS alone group receiving TAU will be recruited as a clinical control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Participants with a confirmed diagnosis of MDD receiving TAU (No Intervention): Eligible and consenting patients will be assigned 1:1 to receive either FMT from a healthy donor or continuing on their usual medication for MDD, i.e., treatment as usual (TAU). This arm will continue to receive their usual anti-depressant.
- Participants with a confirmed diagnosis MDD who will receive FMT + TAU (Active Comparator): Eligible and consenting patients will be assigned 1:1 to receive either FMT from a healthy donor or continuing on their usual medication for MDD, i.e., treatment as usual (TAU). This arm will be assigned to receive FMT provided by healthy donors.
  Interventions: Biological: Fecal Microbiota Transplantation
- Participants with a confirmed diagnosis of MDD + IBS assigned to continue with TAU (No Intervention)
- Participants with a confirmed diagnosis of MDD + IBS assigned to receive FMT + TAU (Active Comparator)
  Interventions: Biological: Fecal Microbiota Transplantation
- Participants with a confirmed diagnosis IBS only receiving TAU (No Intervention)
- Healthy Controls (No Intervention): Data from healthy comparison (HC) participants will be drawn from another completed research study. Healthy comparison participants who will best match the patient population enrolled in the current trial and who consented to data sharing will be selected.

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — FMT is a technique in which intestinal microbiota are transferred from a healthy screened donor to a patient, with the goal being to introduce or restore a stable microbial community in the gut.
  Other Names: FMT
  Arms: Participants with a confirmed diagnosis MDD who will receive FMT + TAU; Participants with a confirmed diagnosis of MDD + IBS assigned to receive FMT + TAU

SUMMARY:
This study is a phase 2/3 open-label controlled trial (CT) in which adults with Major Depressive Disorder (MDD) and adults who have MDD plus comorbid Inflammatory Bowel Syndrome (IBS) will be assigned to either receive oral Fecal Microbiota Transplantation (FMT) or to continue with the treatment they are currently receiving in a Treatment As Usual (TAU) arm. An IBS alone group receiving TAU will be recruited as a clinical control group.

The primary goals of this study are to determine effectiveness, safety and tolerability of oral FMT in adults with MDD and in MDD who have comorbid IBS. Additional goals are to characterize patterns and progressions of cognitive and neural correlates associated with MDD and with MDD + IBS and to determine if they improve with FMT. It is known that both, individuals with MDD and those with MDD and IBS show cognitive alterations as well as changes in neural structures, but this study is designed to see if those are changed with treatment response to FMT."

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-60 years of age:

   Participants should be at least 18 years old and not older than 60 years at the day of screening
2. Have a primary diagnosis of MDD as assessed/confirmed by the M.I.N.I. International Neuropsychiatric Interview (MINI)
3. Have had a well-documented inadequate response to at least 2 approved antidepressants
4. A MADRS score of ≥ 19 at screening and visit 2a
5. Have a comorbid diagnosis of IBS. IBS patients can include any of the following: diarrhea predominant IBS (IBS-D), constipation predominant IBS (IBS-C), IBS with mixed bowel habits (IBS-M), or unclassified with IBS (IBS-U) as confirmed by the referring doctor using ROME III criteria
6. Moderate-to-severe IBS symptoms, as indicated by a score of ≥175 on the IBS Severity Scoring System (IBS-SSS)

Exclusion Criteria:

1. Participant meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5)[1] Criteria for the following conditions according to the M.I.N.I:

   1. Substance Use Disorder within the last 3 months. *(Criteria should include Alcohol and non-alcohol substances except Cannabis)
   2. Moderate or severe substance use disorder for Cannabis use the last 3 months
   3. Active Anorexia Nervosa or Bulimia nervosa
   4. Schizophrenia, schizoaffective or bipolar disorder
   5. Active suicidality
2. Regular intake of non-steroidal anti-inflammatory drugs, antibiotics, or iron supplements for medical purposes in the three (3) months prior to study entry
3. Use of prebiotics or probiotics for medical purposes for more than two (2) weeks within the last three (3) months
4. Conditions causing immunosuppression
5. Women who are breastfeeding, pregnant or seeking to get pregnant during the course of this study. Not using an acceptable method of birth control (implants, injectable, combined oral contraceptives, IUDs, sexual abstinence or a vasectomized partner)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline to week 13
  a 10-item questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. This will be used to evaluate the effectiveness of adjunct oral FMT as compared to TAU with currently accepted approved therapy for MDD.
  The MADRS overall score ranges from 0 to 60. Each item yields a score of 0 to 6 and Higher MADRS score indicates more severe depression
IBS Symptom Severity Scale (IBS-SSS) | Baseline to week 13
  The IBS-SSS is a 5-item questionnaire that is used to assess the severity and frequency of abdominal pain, severity of abdominal distention, dissatisfaction with bowel habits, and interference with quality of life over the past 10 days.
  Scores on the IBS-SSS can range from 0 to 500 with higher scores indicating more severe symptoms. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) IBS.

SECONDARY OUTCOMES:
Toronto Side Effect Scale (TSES) | Baseline to Week 13
  The TSES is a 32-item instrument that is designed to establish incidence, frequency, and severity of CNS, GI, and sexual side effects. For each side effect, frequency and severity are measured on a 5-point scale. intensity is measured by multiplying frequency and severity.
IBS specific Quality of Life (IBS-QoL) | Baseline to Week 13
  is a self-report 34-item instrument used to assess the impact of IBS and its treatment. used to examine GI tolerability in patients with IBS.
  The individual responses to the 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
nuclear magnetic resonance (NMR) spectrometry | Baseline to Week 13
  To assess the effect of FMT on microbiome profile (community structure and functional metagenome).

OTHER OUTCOMES:
structural and functional neuroimaging | Baseline to week 13
  fMRI to examine brain imaging changes in response to FMT

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Taylor, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, TRW building, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Association, A.P., Diagnostic and Statistical Manual of Mental Disorders. 5th Edition ed. 2013, Arlington, VA: American Psychiatric Publishing.
- [Background] Moussavi S, Chatterji S, Verdes E, Tandon A, Patel V, Ustun B. Depression, chronic diseases, and decrements in health: results from the World Health Surveys. Lancet. 2007 Sep 8;370(9590):851-8. doi: 10.1016/S0140-6736(07)61415-9. PMID 17826170
- [Background] Parikh SV, Segal ZV, Grigoriadis S, Ravindran AV, Kennedy SH, Lam RW, Patten SB; Canadian Network for Mood and Anxiety Treatments (CANMAT). Canadian Network for Mood and Anxiety Treatments (CANMAT) clinical guidelines for the management of major depressive disorder in adults. II. Psychotherapy alone or in combination with antidepressant medication. J Affect Disord. 2009 Oct;117 Suppl 1:S15-25. doi: 10.1016/j.jad.2009.06.042. Epub 2009 Aug 13. PMID 19682749
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Colom F, Vieta E, Martinez-Aran A, Reinares M, Benabarre A, Gasto C. Clinical factors associated with treatment noncompliance in euthymic bipolar patients. J Clin Psychiatry. 2000 Aug;61(8):549-55. doi: 10.4088/jcp.v61n0802. PMID 10982196
- [Background] Taylor VH, McIntyre RS, Remington G, Levitan RD, Stonehocker B, Sharma AM. Beyond pharmacotherapy: understanding the links between obesity and chronic mental illness. Can J Psychiatry. 2012 Jan;57(1):5-12. doi: 10.1177/070674371205700103. PMID 22296962
- [Background] Whitehead WE, Crowell MD. Psychologic considerations in the irritable bowel syndrome. Gastroenterol Clin North Am. 1991 Jun;20(2):249-67. PMID 2066151
- [Background] Neufeld KM, Kang N, Bienenstock J, Foster JA. Reduced anxiety-like behavior and central neurochemical change in germ-free mice. Neurogastroenterol Motil. 2011 Mar;23(3):255-64, e119. doi: 10.1111/j.1365-2982.2010.01620.x. Epub 2010 Nov 5. PMID 21054680
- [Background] Lyte M, Li W, Opitz N, Gaykema RP, Goehler LE. Induction of anxiety-like behavior in mice during the initial stages of infection with the agent of murine colonic hyperplasia Citrobacter rodentium. Physiol Behav. 2006 Oct 30;89(3):350-7. doi: 10.1016/j.physbeh.2006.06.019. Epub 2006 Aug 2. PMID 16887154
- [Background] Bravo JA, Forsythe P, Chew MV, Escaravage E, Savignac HM, Dinan TG, Bienenstock J, Cryan JF. Ingestion of Lactobacillus strain regulates emotional behavior and central GABA receptor expression in a mouse via the vagus nerve. Proc Natl Acad Sci U S A. 2011 Sep 20;108(38):16050-5. doi: 10.1073/pnas.1102999108. Epub 2011 Aug 29. PMID 21876150
- [Background] Lyte, M., Microbial endocrinology and nutrition: A perspective on new mechanisms by which diet can influence gut-to-brain communication. PharmaNutrition, 2013. 1(1): p. 35-39. https://doi.org/10.1016/j.phanu.2012.11.002
- [Background] De Palma G, Lynch MD, Lu J, Dang VT, Deng Y, Jury J, Umeh G, Miranda PM, Pigrau Pastor M, Sidani S, Pinto-Sanchez MI, Philip V, McLean PG, Hagelsieb MG, Surette MG, Bergonzelli GE, Verdu EF, Britz-McKibbin P, Neufeld JD, Collins SM, Bercik P. Transplantation of fecal microbiota from patients with irritable bowel syndrome alters gut function and behavior in recipient mice. Sci Transl Med. 2017 Mar 1;9(379):eaaf6397. doi: 10.1126/scitranslmed.aaf6397. PMID 28251905
- [Background] Kelly JR, Borre Y, O' Brien C, Patterson E, El Aidy S, Deane J, Kennedy PJ, Beers S, Scott K, Moloney G, Hoban AE, Scott L, Fitzgerald P, Ross P, Stanton C, Clarke G, Cryan JF, Dinan TG. Transferring the blues: Depression-associated gut microbiota induces neurobehavioural changes in the rat. J Psychiatr Res. 2016 Nov;82:109-18. doi: 10.1016/j.jpsychires.2016.07.019. Epub 2016 Jul 25. PMID 27491067
- [Background] Kurokawa S, Kishimoto T, Mizuno S, Masaoka T, Naganuma M, Liang KC, Kitazawa M, Nakashima M, Shindo C, Suda W, Hattori M, Kanai T, Mimura M. The effect of fecal microbiota transplantation on psychiatric symptoms among patients with irritable bowel syndrome, functional diarrhea and functional constipation: An open-label observational study. J Affect Disord. 2018 Aug 1;235:506-512. doi: 10.1016/j.jad.2018.04.038. Epub 2018 Apr 12. PMID 29684865
- [Background] Duan R, Zhu S, Wang B, Duan L. Alterations of Gut Microbiota in Patients With Irritable Bowel Syndrome Based on 16S rRNA-Targeted Sequencing: A Systematic Review. Clin Transl Gastroenterol. 2019 Feb;10(2):e00012. doi: 10.14309/ctg.0000000000000012. PMID 30829919
- [Background] Fond G, Loundou A, Hamdani N, Boukouaci W, Dargel A, Oliveira J, Roger M, Tamouza R, Leboyer M, Boyer L. Anxiety and depression comorbidities in irritable bowel syndrome (IBS): a systematic review and meta-analysis. Eur Arch Psychiatry Clin Neurosci. 2014 Dec;264(8):651-60. doi: 10.1007/s00406-014-0502-z. Epub 2014 Apr 6. PMID 24705634
- [Background] Luna RA, Foster JA. Gut brain axis: diet microbiota interactions and implications for modulation of anxiety and depression. Curr Opin Biotechnol. 2015 Apr;32:35-41. doi: 10.1016/j.copbio.2014.10.007. Epub 2014 Nov 21. PMID 25448230
- [Background] Camilleri M. Probiotics and irritable bowel syndrome: rationale, putative mechanisms, and evidence of clinical efficacy. J Clin Gastroenterol. 2006 Mar;40(3):264-9. doi: 10.1097/00004836-200603000-00020. PMID 16633134
- [Background] Desbonnet L, Garrett L, Clarke G, Bienenstock J, Dinan TG. The probiotic Bifidobacteria infantis: An assessment of potential antidepressant properties in the rat. J Psychiatr Res. 2008 Dec;43(2):164-74. doi: 10.1016/j.jpsychires.2008.03.009. Epub 2008 May 5. PMID 18456279
- [Background] Eutamene H, Bueno L. Role of probiotics in correcting abnormalities of colonic flora induced by stress. Gut. 2007 Nov;56(11):1495-7. doi: 10.1136/gut.2007.124040. PMID 17938427
- [Background] Gareau MG, Jury J, MacQueen G, Sherman PM, Perdue MH. Probiotic treatment of rat pups normalises corticosterone release and ameliorates colonic dysfunction induced by maternal separation. Gut. 2007 Nov;56(11):1522-8. doi: 10.1136/gut.2006.117176. Epub 2007 Mar 5. PMID 17339238
- [Background] Sullivan A, Nord CE. Probiotics and gastrointestinal diseases. J Intern Med. 2005 Jan;257(1):78-92. doi: 10.1111/j.1365-2796.2004.01410.x. PMID 15606379
- [Background] Girard SA, Bah TM, Kaloustian S, Lada-Moldovan L, Rondeau I, Tompkins TA, Godbout R, Rousseau G. Lactobacillus helveticus and Bifidobacterium longum taken in combination reduce the apoptosis propensity in the limbic system after myocardial infarction in a rat model. Br J Nutr. 2009 Nov;102(10):1420-5. doi: 10.1017/S0007114509990766. Epub 2009 Jun 29. PMID 19563693
- [Background] Logan AC, Katzman M. Major depressive disorder: probiotics may be an adjuvant therapy. Med Hypotheses. 2005;64(3):533-8. doi: 10.1016/j.mehy.2004.08.019. PMID 15617861
- [Background] Rao AV, Bested AC, Beaulne TM, Katzman MA, Iorio C, Berardi JM, Logan AC. A randomized, double-blind, placebo-controlled pilot study of a probiotic in emotional symptoms of chronic fatigue syndrome. Gut Pathog. 2009 Mar 19;1(1):6. doi: 10.1186/1757-4749-1-6. PMID 19338686
- [Background] Messaoudi M, Lalonde R, Violle N, Javelot H, Desor D, Nejdi A, Bisson JF, Rougeot C, Pichelin M, Cazaubiel M, Cazaubiel JM. Assessment of psychotropic-like properties of a probiotic formulation (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175) in rats and human subjects. Br J Nutr. 2011 Mar;105(5):755-64. doi: 10.1017/S0007114510004319. Epub 2010 Oct 26. PMID 20974015
- [Background] Dickerson FB, Stallings C, Origoni A, Katsafanas E, Savage CL, Schweinfurth LA, Goga J, Khushalani S, Yolken RH. Effect of probiotic supplementation on schizophrenia symptoms and association with gastrointestinal functioning: a randomized, placebo-controlled trial. Prim Care Companion CNS Disord. 2014;16(1):PCC.13m01579. doi: 10.4088/PCC.13m01579. Epub 2014 Feb 13. PMID 24940526
- [Background] Dale HF, Rasmussen SH, Asiller OO, Lied GA. Probiotics in Irritable Bowel Syndrome: An Up-to-Date Systematic Review. Nutrients. 2019 Sep 2;11(9):2048. doi: 10.3390/nu11092048. PMID 31480656
- [Background] Majeed M, Nagabhushanam K, Natarajan S, Sivakumar A, Ali F, Pande A, Majeed S, Karri SK. Bacillus coagulans MTCC 5856 supplementation in the management of diarrhea predominant Irritable Bowel Syndrome: a double blind randomized placebo controlled pilot clinical study. Nutr J. 2016 Feb 27;15:21. doi: 10.1186/s12937-016-0140-6. PMID 26922379
- [Background] Ishaque SM, Khosruzzaman SM, Ahmed DS, Sah MP. A randomized placebo-controlled clinical trial of a multi-strain probiotic formulation (Bio-Kult(R)) in the management of diarrhea-predominant irritable bowel syndrome. BMC Gastroenterol. 2018 May 25;18(1):71. doi: 10.1186/s12876-018-0788-9. PMID 29801486
- [Background] Jafari E, Vahedi H, Merat S, Momtahen S, Riahi A. Therapeutic effects, tolerability and safety of a multi-strain probiotic in Iranian adults with irritable bowel syndrome and bloating. Arch Iran Med. 2014 Jul;17(7):466-70. PMID 24979556
- [Background] Mezzasalma V, Manfrini E, Ferri E, Sandionigi A, La Ferla B, Schiano I, Michelotti A, Nobile V, Labra M, Di Gennaro P. A Randomized, Double-Blind, Placebo-Controlled Trial: The Efficacy of Multispecies Probiotic Supplementation in Alleviating Symptoms of Irritable Bowel Syndrome Associated with Constipation. Biomed Res Int. 2016;2016:4740907. doi: 10.1155/2016/4740907. Epub 2016 Aug 9. PMID 27595104
- [Background] Sisson G, Ayis S, Sherwood RA, Bjarnason I. Randomised clinical trial: A liquid multi-strain probiotic vs. placebo in the irritable bowel syndrome--a 12 week double-blind study. Aliment Pharmacol Ther. 2014 Jul;40(1):51-62. doi: 10.1111/apt.12787. Epub 2014 May 11. PMID 24815298
- [Background] Staudacher HM, Lomer MCE, Farquharson FM, Louis P, Fava F, Franciosi E, Scholz M, Tuohy KM, Lindsay JO, Irving PM, Whelan K. A Diet Low in FODMAPs Reduces Symptoms in Patients With Irritable Bowel Syndrome and A Probiotic Restores Bifidobacterium Species: A Randomized Controlled Trial. Gastroenterology. 2017 Oct;153(4):936-947. doi: 10.1053/j.gastro.2017.06.010. Epub 2017 Jun 15. PMID 28625832
- [Background] Wong RK, Yang C, Song GH, Wong J, Ho KY. Melatonin regulation as a possible mechanism for probiotic (VSL#3) in irritable bowel syndrome: a randomized double-blinded placebo study. Dig Dis Sci. 2015 Jan;60(1):186-94. doi: 10.1007/s10620-014-3299-8. Epub 2014 Aug 5. PMID 25092036
- [Background] Hod K, Sperber AD, Ron Y, Boaz M, Dickman R, Berliner S, Halpern Z, Maharshak N, Dekel R. A double-blind, placebo-controlled study to assess the effect of a probiotic mixture on symptoms and inflammatory markers in women with diarrhea-predominant IBS. Neurogastroenterol Motil. 2017 Jul;29(7). doi: 10.1111/nmo.13037. Epub 2017 Mar 8. PMID 28271623
- [Background] Ludidi S, Jonkers DM, Koning CJ, Kruimel JW, Mulder L, van der Vaart IB, Conchillo JM, Masclee AA. Randomized clinical trial on the effect of a multispecies probiotic on visceroperception in hypersensitive IBS patients. Neurogastroenterol Motil. 2014 May;26(5):705-14. doi: 10.1111/nmo.12320. Epub 2014 Mar 4. PMID 24588932
- [Background] EISEMAN B, SILEN W, BASCOM GS, KAUVAR AJ. Fecal enema as an adjunct in the treatment of pseudomembranous enterocolitis. Surgery. 1958 Nov;44(5):854-9. No abstract available. PMID 13592638
- [Background] Health Canada, Guidance Document: Fecal Microbiota Therapy Used in the Treatment of Clostridium difficile Infection Not Responsive to Conventional Therapies. 2015: Ottawa
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290
- [Background] Colman RJ, Rubin DT. Fecal microbiota transplantation as therapy for inflammatory bowel disease: a systematic review and meta-analysis. J Crohns Colitis. 2014 Dec;8(12):1569-81. doi: 10.1016/j.crohns.2014.08.006. Epub 2014 Sep 13. PMID 25223604
- [Background] Zoller V, Laguna AL, Prazeres Da Costa O, Buch T, Goke B, Storr M. [Fecal microbiota transfer (FMT) in a patient with refractory irritable bowel syndrome]. Dtsch Med Wochenschr. 2015 Aug;140(16):1232-6. doi: 10.1055/s-0041-103798. Epub 2015 Aug 11. German. PMID 26261935
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Background] Xu MQ, Cao HL, Wang WQ, Wang S, Cao XC, Yan F, Wang BM. Fecal microbiota transplantation broadening its application beyond intestinal disorders. World J Gastroenterol. 2015 Jan 7;21(1):102-11. doi: 10.3748/wjg.v21.i1.102. PMID 25574083
- [Background] Aroniadis OC, Brandt LJ. Fecal microbiota transplantation: past, present and future. Curr Opin Gastroenterol. 2013 Jan;29(1):79-84. doi: 10.1097/MOG.0b013e32835a4b3e. PMID 23041678
- [Background] Fremont M, Coomans D, Massart S, De Meirleir K. High-throughput 16S rRNA gene sequencing reveals alterations of intestinal microbiota in myalgic encephalomyelitis/chronic fatigue syndrome patients. Anaerobe. 2013 Aug;22:50-6. doi: 10.1016/j.anaerobe.2013.06.002. Epub 2013 Jun 19. PMID 23791918
- [Background] Ananthaswamy, A., Faecal transplant eases symptoms of Parkinson's disease. New Scientist, 2011. 209(2796): p. 8-9 . https://doi.org/10.1016/S0262-4079(11)60124-3
- [Background] Borody, T.J., et al., Fecal microbiota transplantation (FMT) in multiple sclerosis (MS) [abstract]. Am J Gastroenterol, 2011. 106: p. S352 . https://journals.lww.com/ajg/fulltext/2011/10002/fecal_microbiota_transplantation__fmt__in_multiple.942.aspx
- [Background] Diaz Heijtz R, Wang S, Anuar F, Qian Y, Bjorkholm B, Samuelsson A, Hibberd ML, Forssberg H, Pettersson S. Normal gut microbiota modulates brain development and behavior. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3047-52. doi: 10.1073/pnas.1010529108. Epub 2011 Jan 31. PMID 21282636
- [Background] Goehler LE, Gaykema RP, Opitz N, Reddaway R, Badr N, Lyte M. Activation in vagal afferents and central autonomic pathways: early responses to intestinal infection with Campylobacter jejuni. Brain Behav Immun. 2005 Jul;19(4):334-44. doi: 10.1016/j.bbi.2004.09.002. PMID 15944073
- [Background] Bangsgaard Bendtsen KM, Krych L, Sorensen DB, Pang W, Nielsen DS, Josefsen K, Hansen LH, Sorensen SJ, Hansen AK. Gut microbiota composition is correlated to grid floor induced stress and behavior in the BALB/c mouse. PLoS One. 2012;7(10):e46231. doi: 10.1371/journal.pone.0046231. Epub 2012 Oct 2. PMID 23056268
- [Background] Naseribafrouei A, Hestad K, Avershina E, Sekelja M, Linlokken A, Wilson R, Rudi K. Correlation between the human fecal microbiota and depression. Neurogastroenterol Motil. 2014 Aug;26(8):1155-62. doi: 10.1111/nmo.12378. Epub 2014 Jun 1. PMID 24888394
- [Background] Jiang H, Ling Z, Zhang Y, Mao H, Ma Z, Yin Y, Wang W, Tang W, Tan Z, Shi J, Li L, Ruan B. Altered fecal microbiota composition in patients with major depressive disorder. Brain Behav Immun. 2015 Aug;48:186-94. doi: 10.1016/j.bbi.2015.03.016. Epub 2015 Apr 13. PMID 25882912
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Williams JB, Kobak KA. Development and reliability of a structured interview guide for the Montgomery Asberg Depression Rating Scale (SIGMA). Br J Psychiatry. 2008 Jan;192(1):52-8. doi: 10.1192/bjp.bp.106.032532. PMID 18174510
- [Background] Vanderkooy JD, Kennedy SH, Bagby RM. Antidepressant side effects in depression patients treated in a naturalistic setting: a study of bupropion, moclobemide, paroxetine, sertraline, and venlafaxine. Can J Psychiatry. 2002 Mar;47(2):174-80. doi: 10.1177/070674370204700208. PMID 11926080
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Rossen NG, MacDonald JK, de Vries EM, D'Haens GR, de Vos WM, Zoetendal EG, Ponsioen CY. Fecal microbiota transplantation as novel therapy in gastroenterology: A systematic review. World J Gastroenterol. 2015 May 7;21(17):5359-71. doi: 10.3748/wjg.v21.i17.5359. PMID 25954111
- [Background] Hamilton MJ, Weingarden AR, Unno T, Khoruts A, Sadowsky MJ. High-throughput DNA sequence analysis reveals stable engraftment of gut microbiota following transplantation of previously frozen fecal bacteria. Gut Microbes. 2013 Mar-Apr;4(2):125-35. doi: 10.4161/gmic.23571. Epub 2013 Jan 18. PMID 23333862
- [Background] Blais MA, Malone JC, Stein MB, Slavin-Mulford J, O'Keefe SM, Renna M, Sinclair SJ. Treatment as usual (TAU) for depression: a comparison of psychotherapy, pharmacotherapy, and combined treatment at a large academic medical center. Psychotherapy (Chic). 2013 Mar;50(1):110-8. doi: 10.1037/a0031385. PMID 23505987
- [Background] Patrick DL, Drossman DA, Frederick IO, DiCesare J, Puder KL. Quality of life in persons with irritable bowel syndrome: development and validation of a new measure. Dig Dis Sci. 1998 Feb;43(2):400-11. doi: 10.1023/a:1018831127942. PMID 9512138
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Calabrese JR, Bowden CL, Sachs GS, Ascher JA, Monaghan E, Rudd GD. A double-blind placebo-controlled study of lamotrigine monotherapy in outpatients with bipolar I depression. Lamictal 602 Study Group. J Clin Psychiatry. 1999 Feb;60(2):79-88. doi: 10.4088/jcp.v60n0203. PMID 10084633
- [Background] Julious, S.A., Sample Sizes for Clinical Trials. 2009: Chapman and Hall/CRC. 328 Pages.
- [Background] Shein-Chung Chow, J.S., Hansheng Wang, Sample Size Calculations in Clinical Research. 2nd ed. International Statistical Review. Vol. 76. 2008. 301-302.
- [Background] Dear BF, Titov N, Sunderland M, McMillan D, Anderson T, Lorian C, Robinson E. Psychometric comparison of the generalized anxiety disorder scale-7 and the Penn State Worry Questionnaire for measuring response during treatment of generalised anxiety disorder. Cogn Behav Ther. 2011;40(3):216-27. doi: 10.1080/16506073.2011.582138. Epub 2011 Jul 20. PMID 21770844
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Iverson GL, Brooks BL, Young AH. Identifying neurocognitive impairment in depression using computerized testing. Appl Neuropsychol. 2009 Oct;16(4):254-61. doi: 10.1080/09084280903297594. PMID 20183180
- [Background] Kwan ML, Kushi LH, Song J, Timperi AW, Boynton AM, Johnson KM, Standley J, Kristal AR. A practical method for collecting food record data in a prospective cohort study of breast cancer survivors. Am J Epidemiol. 2010 Dec 1;172(11):1315-23. doi: 10.1093/aje/kwq284. Epub 2010 Oct 11. PMID 20937633
- [Background] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603
- [Background] Ye Y. Identification and Quantification of Abundant Species from Pyrosequences of 16S rRNA by Consensus Alignment. Proceedings (IEEE Int Conf Bioinformatics Biomed). 2011 Feb 4;2010:153-157. doi: 10.1109/BIBM.2010.5706555. PMID 22102981
- [Background] Wang Q, Garrity GM, Tiedje JM, Cole JR. Naive Bayesian classifier for rapid assignment of rRNA sequences into the new bacterial taxonomy. Appl Environ Microbiol. 2007 Aug;73(16):5261-7. doi: 10.1128/AEM.00062-07. Epub 2007 Jun 22. PMID 17586664
- [Background] McDonald D, Price MN, Goodrich J, Nawrocki EP, DeSantis TZ, Probst A, Andersen GL, Knight R, Hugenholtz P. An improved Greengenes taxonomy with explicit ranks for ecological and evolutionary analyses of bacteria and archaea. ISME J. 2012 Mar;6(3):610-8. doi: 10.1038/ismej.2011.139. Epub 2011 Dec 1. PMID 22134646
- [Background] DeSantis TZ, Hugenholtz P, Larsen N, Rojas M, Brodie EL, Keller K, Huber T, Dalevi D, Hu P, Andersen GL. Greengenes, a chimera-checked 16S rRNA gene database and workbench compatible with ARB. Appl Environ Microbiol. 2006 Jul;72(7):5069-72. doi: 10.1128/AEM.03006-05. PMID 16820507
- [Background] Lozupone C, Lladser ME, Knights D, Stombaugh J, Knight R. UniFrac: an effective distance metric for microbial community comparison. ISME J. 2011 Feb;5(2):169-72. doi: 10.1038/ismej.2010.133. Epub 2010 Sep 9. No abstract available. PMID 20827291
- [Background] Caporaso JG, Kuczynski J, Stombaugh J, Bittinger K, Bushman FD, Costello EK, Fierer N, Pena AG, Goodrich JK, Gordon JI, Huttley GA, Kelley ST, Knights D, Koenig JE, Ley RE, Lozupone CA, McDonald D, Muegge BD, Pirrung M, Reeder J, Sevinsky JR, Turnbaugh PJ, Walters WA, Widmann J, Yatsunenko T, Zaneveld J, Knight R. QIIME allows analysis of high-throughput community sequencing data. Nat Methods. 2010 May;7(5):335-6. doi: 10.1038/nmeth.f.303. Epub 2010 Apr 11. No abstract available. PMID 20383131
- [Background] McMurdie PJ, Holmes S. Phyloseq: a bioconductor package for handling and analysis of high-throughput phylogenetic sequence data. Pac Symp Biocomput. 2012:235-46. PMID 22174279
- [Background] Le Gall G, Noor SO, Ridgway K, Scovell L, Jamieson C, Johnson IT, Colquhoun IJ, Kemsley EK, Narbad A. Metabolomics of fecal extracts detects altered metabolic activity of gut microbiota in ulcerative colitis and irritable bowel syndrome. J Proteome Res. 2011 Sep 2;10(9):4208-18. doi: 10.1021/pr2003598. Epub 2011 Aug 8. PMID 21761941
- [Background] Psychogios N, Hau DD, Peng J, Guo AC, Mandal R, Bouatra S, Sinelnikov I, Krishnamurthy R, Eisner R, Gautam B, Young N, Xia J, Knox C, Dong E, Huang P, Hollander Z, Pedersen TL, Smith SR, Bamforth F, Greiner R, McManus B, Newman JW, Goodfriend T, Wishart DS. The human serum metabolome. PLoS One. 2011 Feb 16;6(2):e16957. doi: 10.1371/journal.pone.0016957. PMID 21359215
- [Background] DeMets DL, Lan KK. Interim analysis: the alpha spending function approach. Stat Med. 1994 Jul 15-30;13(13-14):1341-52; discussion 1353-6. doi: 10.1002/sim.4780131308. PMID 7973215